CLINICAL TRIAL: NCT06148649
Title: A Phase 2, Multicenter, Randomised, Paralleled, Placebo-controlled (Double-blind) and Active Drug-controlled (Open) Study to Investigate Efficacy and Safety of HEC88473 Injection in Subjects With Type 2 Diabetes Mellitus
Brief Title: Phase 2 Study of HEC88473 Injection in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dongguan HEC Biopharmaceutical R&D Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC88473-DM-201
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- HEC88473 dose1 (Experimental): T2DM subjects, receiving a weekly dose of HEC88473 dose1
  Interventions: Drug: HEC88473, Placebo, Dulaglutide
- HEC88473 dose2 (Experimental): T2DM subjects, receiving a weekly dose of HEC88473 dose2
  Interventions: Drug: HEC88473, Placebo, Dulaglutide
- HEC88473 dose3 (Experimental): T2DM subjects, receiving a weekly dose of HEC88473 dose3
  Interventions: Drug: HEC88473, Placebo, Dulaglutide
- Placebo (Placebo Comparator): T2DM subjects, receiving a weekly dose of placebo
  Interventions: Drug: HEC88473, Placebo, Dulaglutide
- Dulaglutide (Active Comparator): T2DM subjects, receiving a weekly dose of dulaglutide
  Interventions: Drug: HEC88473, Placebo, Dulaglutide

INTERVENTIONS:
Drug: HEC88473, Placebo, Dulaglutide — T2DM subjects, receiving a weekly dose of HEC88473, placebo or dulaglutide.

SUMMARY:
This is a multicenter, randomized, parallel, placebo- and active comparator-controlled phase 2 trial to evaluate the efficacy, safety, pharmacokinetics and immunogenicity in subjects with T2DM.

Patients treated with diet and exercise alone, or in combination with stable metformin monotherapy (≥1500 mg/day or maximum tolerated dose ≥1000 mg/ day.), will be enrolled. Approximately 225 participants will be randomized. The study includes four stages: screening period (up to 2 weeks), lead-in period (2 weeks), treatment period (12 weeks) and safety follow-up period (3 weeks after treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 to 75 years of age, inclusive.
2. Have T2DM for at least 3 months before screening based on the disease diagnostic criteria (WHO 1999).
3. Have an HbA1c value of ≥7.5% and ≤10.5%, fasting blood-glucose ≤13.9 mmoL/L, at screening and visit 3.

Exclusion Criteria:

1. Have type 1 diabetes mellitus.
2. Have had ≥1 episode of severe hypoglycemia within 6 months before screening, or history of recurrent hypoglycemia (history of hypoglycemia more than 3 times in 3 months).
3. Have acute or chronic hepatitis, signs and symptoms of any other liver disease other than nonalcoholic fatty liver disease (NAFLD), or alanine aminotransferase (ALT) level >2.5 times the upper limit of the reference range at screening.
4. Have a personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2) at screening.
5. Have serum calcitonin ≥20 ng/L at screening.
6. Fasted triglycerides > 5.7 mmol/L at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline of HbA1c at week 12 | Baseline to week 12
  HbA1c

SECONDARY OUTCOMES:
Change from baseline of weight at week 12 | Baseline to week 12
  weight
Change from baseline of fasting blood-glucose at week 12 | Baseline to week 12
  fasting blood-glucose
Frequency and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline to week 15
  Adverse Events (AEs) and Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Shijiazhuang People's Hospital, Shijiazhuang, Hebei

IPD SHARING:
Plan to Share IPD: No